CLINICAL TRIAL: NCT03044782
Title: Barriers to Healthcare and Quality of Life for Central Centrifugal Cicatricial Alopecia Patients
Brief Title: Barriers to Care and QOL for CCCA Patients
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Assistant Professor, Dermatology, Northwestern University
Other Study IDs: SP070316
Record Dates: First submitted 2016-12-16; First posted 2017-02-07 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Scarring Alopecia; Central Centrifugal Cicatricial Alopecia; Central Centrifugal Scarring Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: 53-Item Survey

SUMMARY:
The purpose of the current project is twofold; first to determine what personal, historical, logistical, and environmental factors preclude women from obtaining medical care for CCCA hair loss. Because damage from CCCA is irreversible, early identification and treatment is paramount to limiting the negative ramifications of the disease. Second, to investigate how CCCA hair loss, a common occurrence in the Black population, can be a significant psychological impediment to lives of affected Black women. Based on previous research on the psychosocial impact of generalized hair loss in Black women, it is fair to consider that CCCA hair loss also leads to problems with self-esteem and participation in daily life activities. This research, the first of its kind, will add to existing knowledge of CCCA by investigating the quality of life and barriers to care of patients with this condition. The goal of this study is to illuminate what stands in the way of secondary and tertiary prevention of CCCA patients and tailor treatment strategies to address their needs. The results of this study will be instrumental in modifying dermatology resident training, adding to existing dermatology management guidelines, and even developing public health advocacy programming.

ELIGIBILITY:
Inclusion Criteria:

* Evaluated in the Northwestern Dermatology Department between October 1, 2015 and September 30, 2017.
* Evaluated by any faculty physician.
* Diagnosed with CCCA.
* Age 18 or older.
* All subjects must have given signed informed consent prior to participation in study.

Exclusion Criteria:

* Non-English speakers (interpreters not available)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with CCCA who have been seen at Northwestern Dermatology between 10/1/15 and 9/30/17.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Quantified Barriers to Care Survey Responses | Duration of study-approximately 2 years
Quantified Quality of Life Survey Responses | Duration of study-approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Kundu, MD, Principal Investigator — Northwestern Department of Dermatology
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dlova NC, Forder M. Central centrifugal cicatricial alopecia: possible familial aetiology in two African families from South Africa. Int J Dermatol. 2012 Nov;51 Suppl 1:17-20, 20-3. doi: 10.1111/j.1365-4632.2012.05557.x. No abstract available. English, French. PMID 23210944
- [Result] Gathers RC, Jankowski M, Eide M, Lim HW. Hair grooming practices and central centrifugal cicatricial alopecia. J Am Acad Dermatol. 2009 Apr;60(4):574-8. doi: 10.1016/j.jaad.2008.10.064. PMID 19293007
- [Result] Gathers RC, Mahan MG. African american women, hair care, and health barriers. J Clin Aesthet Dermatol. 2014 Sep;7(9):26-9. PMID 25276273
- [Result] Halder RM, Grimes PE, McLaurin CI, Kress MA, Kenney JA Jr. Incidence of common dermatoses in a predominantly black dermatologic practice. Cutis. 1983 Oct;32(4):388, 390. PMID 6226496
- [Result] Mkentane K, Maneli M, Khumalo NP, Davids LM, Freedom G. Relaxers damage hair and increase fragility. Int J Dermatol. 2014 Mar;53(3):e200-2. doi: 10.1111/ijd.12283. No abstract available. PMID 24571594
- [Result] Summers P, Kyei A, Bergfeld W. Central centrifugal cicatricial alopecia - an approach to diagnosis and management. Int J Dermatol. 2011 Dec;50(12):1457-64. doi: 10.1111/j.1365-4632.2011.05098.x. PMID 22097988
- [Result] Kyei A, Bergfeld WF, Piliang M, Summers P. Medical and environmental risk factors for the development of central centrifugal cicatricial alopecia: a population study. Arch Dermatol. 2011 Aug;147(8):909-14. doi: 10.1001/archdermatol.2011.66. Epub 2011 Apr 11. PMID 21482861
- [Result] LoPresti P, Papa CM, Kligman AM. Hot comb alopecia. Arch Dermatol. 1968 Sep;98(3):234-8. No abstract available. PMID 5673883
- [Result] Ogunleye TA, McMichael A, Olsen EA. Central centrifugal cicatricial alopecia: what has been achieved, current clues for future research. Dermatol Clin. 2014 Apr;32(2):173-81. doi: 10.1016/j.det.2013.12.005. Epub 2014 Jan 22. PMID 24680004
- [Result] McMichael AJ. Ethnic hair update: past and present. J Am Acad Dermatol. 2003 Jun;48(6 Suppl):S127-33. doi: 10.1067/mjd.2003.278. PMID 12789165
- [Result] Sperling LC, Cowper SE. The histopathology of primary cicatricial alopecia. Semin Cutan Med Surg. 2006 Mar;25(1):41-50. doi: 10.1016/j.sder.2006.01.006. PMID 16616302
- [Result] Sperling LC, Sau P. The follicular degeneration syndrome in black patients. 'Hot comb alopecia' revisited and revised. Arch Dermatol. 1992 Jan;128(1):68-74. PMID 1739290
- [Result] Sperling LC, Solomon AR, Whiting DA. A new look at scarring alopecia. Arch Dermatol. 2000 Feb;136(2):235-42. doi: 10.1001/archderm.136.2.235. No abstract available. PMID 10677100
- [Result] Mukherjee N, Morrell DS, Duvic M, Stewart PW, Goldsmith LA. Attitudes of dermatologists in the southeastern United States regarding treatment of alopecia areata: a cross-sectional survey study. BMC Dermatol. 2009 Nov 12;9:11. doi: 10.1186/1471-5945-9-11. PMID 19909522